CLINICAL TRIAL: NCT06785896
Title: Analysis of the Effect oh the Carriere Motion 3D on Patients With Class II Subdivision : a Retrospective Study
Brief Title: Analysis of the Effect oh the Carriere Motion 3D
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 24Odonto04
Record Dates: First submitted 2024-12-19; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2024-12

CONDITIONS: Angle Class II
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Angle Class II unilateral, treated by carriere motion appliance: This treatment was unilateral, with dental composite bites ramps behind canines
  Interventions: Procedure: Angle Class II unilateral, treated by carriere motion appliance

INTERVENTIONS:
Procedure: Angle Class II unilateral, treated by carriere motion appliance — This treatment was unilateral, with dental composite bites ramps behind canines

SUMMARY:
Class II subdivision malocclusions are common and complex to treat due to their asymmetry. The range of orthodontic correction devices is expanding towards systems that are more comfortable for the patient but may not necessarily have scientific evidence to demonstrate their effectiveness. The aim of this study was therefore to evaluate, for the first time, the effect of a Class II correction device, namely the Carriere Motion 3D (CMA), on patients with a Class II subdivision malocclusion. Method:this retrospective observational study included all patients presenting with a Class II subdivision malocclusion and treated with CMA between July 2018 and November 2023. Before treatment (T0) and after treatment with CMA (T1), orthodontic data from dental molds and lateral cephalometric radiographs (Steiner analysis) were collected and statistically analyzed to assess dentoalveolar as well as skeletal effects of treatment using CMA."

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed their growth and present with a Class II subdivision malocclusion.
* Patients who underwent orthodontic treatment with CMA between 07/11/2018 and 11/22/2023.
* Patients who have a complete orthodontic record allowing for pre- and post-treatment measurements with CMA.

Exclusion Criteria: None

Ages: 28 Years to 47 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consisted of patients treated by Dr. Romain de Papé at his practice in Strasbourg, within the established time frame.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Molar Angle class II correction | Up to 6 months
  Measured between the centro vestibular groove of the maxillar fisrt molar and the mesio vestibulair cusp tip of the mandibular molar in millimeters

SECONDARY OUTCOMES:
Canine Angle class II correction | Up to 6 months
  Measurement performed between the maxillary canine cusp tip and the inter-dental space between the mandibular canine and premolar in millimeters
Extrusion or intrusion | Up to 6 months
  Extrusion or intrusion of the maxillary canines and molars supporting the orthodontic appliance in millimeters
Correction of the Class II canine relationship | Up to 6 months
  Mesured correction of the Class II canine relationship in millimeters
Rotations | Up to 6 months
  Mesured of the Rotations of the molars and canines supporting the CMA in degrees
Inter-incisal variations | Up to 6 months
  Mesure of the variation in the inter-incisal midline discrepancy in millimeters
Arch depth | Up to 6 months
  Mesure of the variation in arch depth in millimeters
Arch width | Up to 6 months
  Mesure of th variation in canine and molar arch width in millimeters
Steiner analysis | Up to 24 months
  A Steiner analysis was performed on the lateral cephalograms, measurements in millimeters on the X-Ray

CONTACTS AND LOCATIONS:
Locations (1):
- CHU NICE, Nice, Alpes Maritimes, France